CLINICAL TRIAL: NCT00910806
Title: A Phase I, Open-label, Single-sequence Drug-drug Interaction Trial to Investigate the Pharmacokinetic Interaction Between Steady-state Nevirapine and Single-dose TMC207 in HIV-1 Infected Subjects.
Brief Title: TMC207-TiDP13-C117: Interaction Study in Human Immunodeficiency Virus-type 1 (HIV-1) Infected Patients With Nevirapine (NVP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015793; NCT00980668 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-06-01 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: TMC207-TiDP13-C117; TMC207-C110; TMC207; drug-drug interaction; Tuberculosis; HIV; nevirapine; open-label; Pharmacokinetics
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — bedaquiline; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TMC207, nevirapine (Experimental)
  Interventions: Drug: TMC207; nevirapine

INTERVENTIONS:
Drug: TMC207; nevirapine

SUMMARY:
The purpose of this Phase I, open-label, single sequence drug-drug interaction trial in human immunodeficiency virus-type 1 infected patients is to investigate the potential interaction between steady-state nevirapine (NVP) 200 mg b.i.d. (twice a day) and a single dose of 400 mg TMC207 and to explore the pharmacokinetics (how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body).

DETAILED DESCRIPTION:
TMC207 is being investigated for the treatment of M. tuberculosis (TB) infection. This is a Phase I, open-label (both participant and investigator know the name of the assigned medication), single-sequence (all participants receive treatments in the same order) drug-drug interaction trial in human immunodeficiency virus - type 1 (HIV-1) infected patients to investigate the potential interaction between steady-state nevirapine (NVP) 200 mg b.i.d. (twice a day) and a single dose of 400 mg TMC207. The study medication will be taken orally. The trial population will consist of 16 patients infected with HIV-1 virus who have not yet been treated for this infection (antiretroviral or ARV naïve) with a medical indication to start ARV therapy and electing to start treatment with NVP plus two nucleos(t)ide reverse transcriptase inhibitors (N(t)RTIs). The primary objective is to evaluate the effect of steady-state NVP 200 mg b.i.d. on the pharmacokinetics of TMC207 and its M2 metabolite after single-dose administration of TMC207 400 mg, in HIV-1 infected patients. The secondary objectives are to evaluate the effect of single-dose TMC207 400 mg on the steady-state plasma concentrations of NVP 200 mg b.i.d. and to evaluate the short-term safety and tolerability of coadministration of single-dose TMC207 and steady-state NVP in HIV-1 infected patients. Prior to starting the NVP-containing regimen, patients will receive a single dose of TMC207 400 mg (Treatment A). At least 2 but no more than 4 weeks later, NVP will be started (in combination with 2 N(t)RTIs) at the recommended dosing regimen (200 mg once daily for 2 weeks followed by 200 mg twice daily). After 4 weeks of NVP at a dose of 200 mg b.i.d., a second single dose of TMC207 400 mg will be administered (Treatment B).Pharmacokinetic profiles over 336 hours will be determined for TMC207 and its N-monodesmethyl metabolite (M2) after administration of TMC207 400 mg alone, and in combination with steady-state NVP. Morning predose concentrations of NVP will be determined at several time points.Safety and tolerability will be evaluated throughout the trial. Adverse events will be recorded at every visit. A blood and urine sample will be taken at screening, day -1, 1, 2 and 15 of treatment A and B and at both follow-up visits. An electrocardiogram will be recorded at screening, twice on day 1 and once on day 2 and 15 of treatment A and B and at the last follow-up visit. Vital signs will be measured at screening, on day 1, 2 and 15 of treatment A and B and at both follow-up visits. A physical examination will be performed at screening, on day -1 of treatment A and B and at both follow-up visits. On day 1 of treatment A and B 400 mg TMC207 (4 tablets) will be taken by mouth in the morning within 10 minutes after completion of the breakfast. At least 2 but no more than 4 weeks after the first single dose of TMC207, NVP will be started [in combination with 2 N(t)RTIs] as 200 mg once daily for 2 weeks followed by 200 mg twice daily, orally. After 4 weeks of NVP at a dose of 200 mg twice daily, a second single dose of TMC207 will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Antiretroviral naïve patients, for whom in the judgment of the investigator, it is appropriate to initiate NVP-containing ARV therapy at least 2 but no more than 4 weeks after the first dose of TMC207, based on the patient's medical condition and taking into account local treatment guidelines for the treatment of HIV-1 infection
* Patient agrees not to start ARV therapy until at least 2 weeks after the first dose of TMC207
* patient agrees not to change NVP and N(t)RTI therapy (including dosages) from the start of NVP treatment at 200 mg b.i.d. until Day 15 of Treatment B, unless this is medically indicated as decided by the treating physician.

Exclusion Criteria:

* Female, except if postmenopausal since more than 2 years, or posthysterectomy, or post-surgical sterilization
* Patient has any currently active AIDS defining illness
* Active tuberculosis
* Known or suspected acute HIV-1 infection
* Currently active or underlying gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, or respiratory disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of steady-state NVP 200 mg twice daily on the pharmacokinetics of TMC207 and its M2 metabolite after single-dose administration of TMC207 400 mg, in HIV-1 infected patients | Pharmacokinetic profiles over 336 hours will be determined for TMC207 and its N-monodesmethyl metabolite (M2) after administration of TMC207 400 mg alone, and in combination with steady-state NVP.

SECONDARY OUTCOMES:
The effect of single-dose TMC207 on the steady-state plasma concentrations of NVP will be evaluated. | This will be determined during 18 days in treatment B
The short-term safety and tolerability of coadministration of single-dose TMC207 and steady-state NVP will be evaluated in HIV-1 infected patients. | This will be determined during 15 days in treatment B

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA
Locations (1):
- George, South Africa

REFERENCES:
- [Derived] Svensson EM, Dooley KE, Karlsson MO. Impact of lopinavir-ritonavir or nevirapine on bedaquiline exposures and potential implications for patients with tuberculosis-HIV coinfection. Antimicrob Agents Chemother. 2014 Nov;58(11):6406-12. doi: 10.1128/AAC.03246-14. Epub 2014 Aug 11. PMID 25114140